CLINICAL TRIAL: NCT04433169
Title: A Prospective, Open-label, Randomized Controlled Clinical Study to Evaluate the Efficacy and Safety of All-trans Retinoic Acid (ATRA) in the Treatment of Patients With Recurrent/Metastatic Adenoid Cystic Carcinoma of the Head and Neck
Brief Title: All-trans Retinoic Acid (ATRA) in the Treatment of Recurrent/Metastatic Adenoid Cystic Carcinoma of the Head and Neck
Acronym: Aplus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020HNRT02
Record Dates: First submitted 2020-06-12; First posted 2020-06-16 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-06

CONDITIONS: Adenoid Cystic Carcinoma of the Head and Neck
MeSH Terms: interventions — Tretinoin; Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): ATRA 20 mg, three times a day (tid), for 28 consecutive days, 28 days per cycle (q4w), 6 planned cycles; combined with the treatment regimen chosen by the investigator since Day 6 of cycle 1.
  Interventions: Drug: All-trans Retinoic Acid
- Control group (Active Comparator): The investigator chooses the treatment regimen based on the following regimens (including but not limited to: 1. VEGFR inhibitor; 2. chemotherapy).
  Interventions: Drug: VEGFR inhibitor; Drug: Chemotherapy

INTERVENTIONS:
Drug: All-trans Retinoic Acid — ATRA 20 mg, three times a day, for 28 consecutive days, 28 days per cycle (q4w), 6 planned cycles
  Other Names: Ailike
  Arms: Experimental group
Drug: VEGFR inhibitor — VEGFR inhibitor
  Arms: Control group
Drug: Chemotherapy — chemotherapy
  Arms: Control group

SUMMARY:
This is a prospective, open-label, randomized controlled clinical intervention study to evaluate the efficacy and safety of all-trans retinoic acid (ATRA) in treating patients with recurrent metastatic adenoid cystic carcinoma of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, male or female; 2. ECOG PS (performance status) score: 0-1; 3. Pathologically or histologically confirmed advanced, recurrent/metastatic ACC, with measurable disease (≥10 mm by spiral CT scan, meeting RECIST 1.1 criteria); 4. Patients with therapeutic indications; 5. Main organ functions normal, i.e., meeting the criteria below:

1. Criteria for routine blood test: (no blood transfusion within 14 days)

   1. HB ≥ 90 g/L;
   2. WBC ≥ 3.5 × 109/L and < 10 × 109/L;
   3. ANC ≥ 1.5 × 109/L;
   4. PLT ≥ 80 × 109/L
2. Criteria for biochemical tests:

   1. BIL < 1.25 × upper limit of normal (ULN)
   2. ALT and AST < 2.5 × ULN; in the presence of metastases to liver, ALT and AST < 5 × ULN;
   3. Serum Cr ≤ 1 × ULN, endogenous creatinine clearance > 50 mL/min (Cockcroft-Gault equation); 5. Subjects who volunteer to participate in this study, sign the informed consent, have good compliance and cooperate in follow-up; 6. Patients who, in the doctor's opinion, can benefit from the treatment.

Exclusion Criteria:

1. Previous or existing concomitant malignancies except cured skin basal cell carcinoma or cervical carcinoma in situ;
2. Coagulation abnormal (INR>1.5, APTT>1.5×ULN), history of gastrointestinal hemorrhage in the past 6 months or bleeding tendency [e.g., presence of active ulcer focus in the stomach, stool occult blood (++), melena and/or hematemesis, hemoptysis in the past 3 months];
3. Confirmed hypersensitivity to ATRA;
4. Grade I and above coronary artery diseases, arrhythmias [including QTc prolongation (males: > 450 ms, females: > 470 ms)] and cardiac dysfunction;
5. Presence of multiple factors affecting oral administration (e.g. dysphagia, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc.);
6. Pregnant or lactating women;
7. History of psychotropic abuse with abstinence failure, or existing mental disorder;
8. Participation in other drug clinical trials within 4 weeks;
9. Other concomitant diseases which seriously jeopardize the patient's safety or prevent the patient from completing the study, as judged by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (CR+PR) | 6 months
  Objective Response Rate as defined by RECIST 1.1 after induction therapy followed by definitive chemoradiation. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective Response (OR) = CR + PR.

SECONDARY OUTCOMES:
Number of Participants With at Least One Grade 3-4 Toxicity | 6 months
  Toxicity will be assessed according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Progression-Free Survival | 6 months
  Time to death or progression defined by imaging of target lesions via CT or MRI scan every 3 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No